CLINICAL TRIAL: NCT05910307
Title: Synovial Sarcoma Registry and Biospecimen Repository
Brief Title: Synovial Sarcoma Registry / Biospecimen Repository
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 23-021012
Record Dates: First submitted 2023-06-01; First posted 2023-06-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Synovial Sarcoma
Keywords: registry; biorepository; sarcoma; oncology; cancer; rare tumor
MeSH Terms: conditions — Sarcoma, Synovial; Sarcoma; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Samples may include tumor tissue and its excipients (DNA, RNA, protein), blood, saliva, and/or buccal swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to collect and store data and samples for future research to attempt to improve outcomes for patients with synovial sarcoma. The future research will involve various types of genetic testing.

Participants will be asked to allow access to medical records and leftover tumor tissue and may be asked to give a blood or saliva sample. Participants will also be asked to completed questionnaires about their medical history and may be contacted every 6 to 12 months for updates for up to 10 years.

DETAILED DESCRIPTION:
This study will enroll patients with a diagnosis of Synovial Sarcoma.

Following consent, demographic, clinical, treatment and outcome data will be collected from an interview and/or online survey. This will include a request for contact information for the subject's treating hospitals/physicians and a release of records request to obtain medical records.

At approximately 6-12 month intervals for up to 10 years after initial diagnosis and/or relapse, subjects and/or their treating hospitals may be contacted to provide updates on treatment and outcomes.

Tumor samples may be collected from residual material obtained during clinically indicated procedures occurring before or after consent to this study. No additional material will be collected or procedures performed solely for the purpose of this study.

Blood may be collected at the participant's local institution at the time of a clinically indicated blood draw and/or saliva or a buccal swab may be collected as a germline sample and for analysis of circulating free DNA (cfDNA) and/or circulating tumor cells (CTCs).

Genetic testing may be performed on tumor and germline samples submitted by subjects. Results will only be returned if deemed clinically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of any age
2. Reported diagnosis of synovial sarcoma
3. Informed consent from subject (aged ≥18 years) or parent/guardian

Exclusion Criteria:

1. Individuals with sarcomas that do not fit the definition of those considered for this registry
2. Individuals who are unwilling to participate
3. Individuals who are unwilling or unable to provide written consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and females of any age with a reported diagnoses of synovial sarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with synovial sarcoma | Up to 10 years
  Number of patients with synovial sarcoma

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Laetsch, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and specimens may be provided to other investigators for additional research use. Identifiable data will only be available to the study team.
Supporting Information: Study Protocol, ICF
Time Frame: Upon request, data can be made available after review by study team.
Access Criteria: The study team will review requests on an individual basis.

REFERENCES:
- See also: Interest Form for Potential Participants — https://redcap.link/synovialsarcomaregistry
- See also: Self-Guided Consent for Potential Participants — https://redcap.link/ssrbconsent
- See also: Study Website — https://www.research.chop.edu/synovial-sarcoma-registry-biospecimen-repository